CLINICAL TRIAL: NCT02303405
Title: Comparing the Effects of Hydroxychloroquine (HCQ) to Pioglitazone in Type 2 Diabetic Patients Failing Maximal Doses of Metformin Plus a Sulfonylurea
Brief Title: Hydroxychloroquine Versus Pioglitazone in Combination Treatment for Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-01-2419
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Results first posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus Type 2 With Hyperglycemia
Keywords: Glucose Control; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Hydroxychloroquine; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxychloroquine (Experimental): Treatment with hydroxychloroquine 400 mg (2 x 200 mg tablets) po once daily x 4 months
  Interventions: Drug: Hydroxychloroquine
- Pioglitazone (Active Comparator): Treatment with pioglitazone 45 mg po (1 tablet) once daily x 4 months
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Hydroxychloroquine — Anti-inflammatory and anti-malarial agent
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: Pioglitazone — Anti-hyperglycemic agent
  Other Names: Actos
  Arms: Pioglitazone

SUMMARY:
A 4-month, randomized, prospective, open-label comparison trial of hydroxychloroquine vs. pioglitazone in type 2 diabetic patients inadequately controlled on maximally tolerated doses of metformin plus a sulfonylurea.

DETAILED DESCRIPTION:
A 4-month, randomized, prospective, open-label comparison trial of 4 months of hydroxychloroquine vs. pioglitazone in type 2 diabetic patients inadequately controlled on maximally tolerated doses of metformin plus a sulfonylurea.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-75, inclusive
* Known type 2 diabetes (diagnosed according to 1997 ADA diagnostic criteria)
* At least 3 months of treatment with maximum tolerated doses of metformin and a sulfonylurea
* Hemoglobin A1c ≥ 7.5% and < 11.0%
* Body mass index (BMI) < 45 kg/m2
* Able to comply with all scheduled visits and requirements of the protocol

Exclusion Criteria:

* Any contraindications to the use of metformin or a sulfonylurea
* Extreme hyperglycemia (FPG ≥ 300 mg/dL), symptoms of polyuria or polydipsia, or Hemoglobin A1c ≥ 11.0%
* Current use of insulin; history or clinical suspicion of type 1 diabetes mellitus
* Symptomatic hypoglycemia occurring at an average frequency > once per day
* Highly erratic dietary schedules, extremely food insecure households, or homelessness that may adversely affect good glycemic control, as judged by the investigators
* Occupations that involve regular operation of motor vehicles or other heavy machinery that may pose a hazard in the event of unanticipated blurred vision
* Known history of Class III or IV heart failure, cardiac arrhythmias, severe peripheral edema, advanced osteoporosis, documented bladder malignancies, or other intolerance to pioglitazone
* Known history of collagen vascular disorders, glucose-6-phosphate dehydrogenase deficiency, hematologic disorders, psoriasis, or any known intolerance to hydroxychloroquine
* Known history of pre-proliferative or proliferative retinopathy, or any clinically significant retinal abnormalities noted on the patient's most recent (i.e., within 1 year) ophthalmologic exam; subjects who have not received their routine annual ophthalmologic surveillance for diabetic retinopathy within the past year must have their annual surveillance performed before screening
* An estimated GFR (by the Modification of Diet in Renal Disease (MDRD) formula) < 45 mL/min, or a history of nephrotic syndrome (defined as a spot urine protein-creatinine ratio of > 3500 mg per g urine creatinine)
* Subjects with active hemoglobin abnormalities that render the Hemoglobin A1c measurement unreliable
* History of any clinically significant hepatic, cardiovascular, infectious, dermatologic, psychiatric, or other major systemic disease that, in the opinion of the investigator, may make the use of pioglitazone or hydroxychloroquine unsafe, or otherwise make the interpretation of the data difficult.
* Female subjects of childbearing potential who are sexually active and not using a reliable form of contraception or do not agree to use a reliable form of contraception. Reliable forms of contraception include systemic contraceptives (oral, implant or injection), diaphragm with spermicide, cervical cap, IUD, or condoms with spermicide.
* Current pregnancy or lactation.
* Subjects who will likely require or initiate therapy with drugs that may interfere with glucose metabolism during the course of the study (e.g., glucocorticoids).
* Subjects who are in another investigational study or have received another investigational medication within 30 days of study entry
* Subjects who are unable or unwilling to give informed consent, comply with all components of the study protocol, attend all scheduled follow-up visits, or present other barriers that would make the implementation of the protocol unusually difficult.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley H Hsia, MD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxychloroquine | Pioglitazone
Started | 15 (Two subjects failed to provide any data after randomization, and were excluded from analyses.) | 7
Completed | 15 (Two subjects failed to provide data at 4 months; last observed data were carried forward.) | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Pioglitazone | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10) | 57 (13) | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latino | 12 | 7 | 19
  Black | 2 | 0 | 2
  Other | 1 | 0 | 1
Diabetes Duration [Mean (Standard Deviation); unit: years] | 5.1 (3.1) | 7.8 (4.3) | 6.0 (3.6)
Weight [Mean (Standard Deviation); unit: kg] | 85.7 (14.3) | 83.7 (18.2) | 85.0 (15.2)
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 8.6 (1.0) | 9.1 (0.7) | 8.7 (0.9)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 179 (53) | 170 (50) | 176 (51)
Body Mass Index [Mean (Standard Deviation); unit: kg per meter squared] | 35.3 (5.7) | 34.1 (5.2) | 34.9 (5.4)
hs-CRP [Mean (Standard Deviation); unit: mg/L] | 6.2 (6.7) | 8.8 (7.2) | 7.0 (6.8)
Leucocyte Count [Mean (Standard Deviation); unit: x 10^9 cells/L] | 8.4 (1.6) | 7.8 (1.4) | 8.2 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: Glycemic control
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
% of hemoglobin | 7.4 (0.9) | 6.3 (0.2)

2. Secondary Outcome: Fasting Plasma Glucose
Description: Fasting glucose level
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
mg/dL | 147 (33) | 105 (21)

3. Secondary Outcome: Percent of Subjects Achieving HbA1c < 7.5%
Description: Percent of subjects achieving a HbA1c level < 7.5%
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
Participants | 10 | 7

4. Secondary Outcome: Weight
Description: Body weight
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
kilograms | 85.4 (14.5) | 87.0 (17.9)

5. Secondary Outcome: Body Mass Index
Description: Body mass index (BMI)
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: kg per square meter
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
kg per square meter | 35.2 (6.0) | 35.5 (5.4)

6. Secondary Outcome: HOMA-IR
Description: Insulin resistance by the HOMA model
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: uU/mL*mg/dL
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
uU/mL*mg/dL | 3.91 (2.92) | 1.48 (0.79)

7. Secondary Outcome: QUICKI
Description: Insulin resistance by the QUICKI model
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: (Log(uU/dL)+Log(mg/dL))^-1
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
(Log(uU/dL)+Log(mg/dL))^-1 | 0.32 (0.03) | 0.38 (0.05)

8. Secondary Outcome: Hs-CRP
Description: Highly-sensitive C-reactive protein (inflammatory marker)
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
mg/L | 4.2 (3.8) | 3.3 (3.7)

9. Secondary Outcome: Leucocyte Count
Description: White cell count (surrogate marker of inflammation)
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: x 10^9 cells/ L
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
x 10^9 cells/ L | 7.7 (1.9) | 6.8 (1.7)

10. Secondary Outcome: Hypoglycemic Events
Description: Number of hypoglycemic events
Time Frame: 4 months
Measure: Number; unit: Events
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
Events | 0 | 6.0

11. Secondary Outcome: Adverse Events
Description: All other adverse events other than hypoglycemia
Time Frame: 4 months
Measure: Number; unit: Events
Arm/Group | Hydroxychloroquine | Pioglitazone
Number analyzed (Participants) | 15 | 7
Events | 0 | 1.0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Hydroxychloroquine | Pioglitazone
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/7
Other Adverse Events (participants affected / at risk) | 0/15 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=15) | Pioglitazone (N=7)
Transient Ischemic Attack (Vascular disorders) | 1 (1) | 0 (0) — Determined as not related to IP
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=15) | Pioglitazone (N=7)
Pedal Edema (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size, Unblinded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT02303405/Prot_SAP_000.pdf